CLINICAL TRIAL: NCT05242432
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate Efficacy, Safety, Reactogenicity, and Immunogenicity of an Ad26.RSV.preF-based Vaccine in Japanese Adults Aged 60 Years and Older, and Safety, Reactogenicity, and Immunogenicity of the Vaccine in Japanese Adults Aged 20 to 59 Years at High-risk of RSV Disease
Brief Title: A Study of Adenovirus Serotype 26.Respiratory Syncytial Virus.Pre-Fusion F (Ad26.RSV.preF)-Based Vaccine for Prevention of Respiratory Syncytial Virus (RSV) Mediated- Lower Respiratory Tract Disease (LRTD) in Japanese Participants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated (Janssen made the strategic decision to discontinue the RSV3007 study. This decision is not based on any safety concerns.)
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109164; VAC18193RSV3007 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Prevention

STUDY DESIGN:
Intervention Model Description: Cohort 1: adults aged 60 years and older Cohort 2: adults aged 20 to 59 years at high-risk of severe RSV disease
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort (C)1 Group (G)1: Adults, 60 years and older (Ad26/protein preF RSV Vaccine) (Experimental): Participants will receive a single intramuscular (IM) injection of Adenovirus Serotype 26.Respiratory Syncytial Virus.Pre-Fusion F (Ad26/protein preF RSV) vaccine on Day 1.
  Interventions: Biological: Ad26/protein preF RSV Vaccine
- C1 G2: Adults, 60 years and older (Placebo) (Placebo Comparator): Participants will receive a single IM injection of matching placebo on Day 1.
  Interventions: Other: Placebo
- C2 G3: Adults Aged 20 to 59 years at High-risk of Severe RSV Disease (Ad26/protein preF RSV Vaccine) (Experimental): Participants will receive a single IM injection of Ad26/protein preF RSV vaccine on Day 1.
  Interventions: Biological: Ad26/protein preF RSV Vaccine
- C2 G4: Adults Aged 20 to 59 years at High-risk of Severe RSV Disease (Placebo) (Placebo Comparator): Participants will receive a single IM injection of matching placebo on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ad26/protein preF RSV Vaccine — Ad26/protein preF RSV vaccine will be administered as an IM injection.
  Other Names: VAC18193
  Arms: C2 G3: Adults Aged 20 to 59 years at High-risk of Severe RSV Disease (Ad26/protein preF RSV Vaccine); Cohort (C)1 Group (G)1: Adults, 60 years and older (Ad26/protein preF RSV Vaccine)
Other: Placebo — Matching Placebo will be administered as an IM injection
  Arms: C1 G2: Adults, 60 years and older (Placebo); C2 G4: Adults Aged 20 to 59 years at High-risk of Severe RSV Disease (Placebo)

SUMMARY:
The purpose of the study is to evaluate the efficacy of study vaccine in the prevention of Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)-confirmed RSV mediated- lower Respiratory Tract Disease (LRTD) over one RSV season when compared to placebo in adults aged 60 years and above and to demonstrate the non-inferiority of the vaccine in high-risk adults aged 20 to 59 years versus in adults aged 60 years and older in terms of humoral immune response.

ELIGIBILITY:
Inclusion Criteria:

For Participants in Cohort 1 only

* Must be greater than or equal to (>=60) years old on the day of signing the informed consent form (ICF) and expected to be available for the duration of the study
* Before randomization, a participant must be postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause); and not intending to conceive by any methods
* Participants may have underlying illnesses such as hypertension, congestive heart failure (CHF), Chronic obstructive pulmonary disease (COPD), type 2 diabetes, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are stable and medically controlled in the judgement of the investigator at the time of vaccination, and these conditions receive routine follow-up by the participant's healthcare provider

For Participants in Cohort 2 only

* Must be aged 20 to 59 years (inclusive) on the day of signing the ICF and expected to be available for the duration of the study
* Has an existing chronic heart or lung condition, without hospitalizations or major medication class change (that is, new or stopped medications) within 30 days prior to screening
* Participant may have other underlying illnesses as long as their symptoms and signs are stable at the time of vaccination, and these conditions receive routine follow-up by the participant's healthcare provider

Exclusion Criteria:

* Has a serious clinically unstable condition like, (example, end-stage renal disease with or without dialysis, clinically unstable cardiac disease), Alzheimer's disease, or any other condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise well-being) or that could prevent or limit the protocol-specified assessments
* History of malignancy within 5 years before screening or revaccination not in the following categories: a. participants with squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix may be enrolled at the discretion of the investigator; b. participants with a history of malignancy within 5 years, which is considered cured with minimal risk of recurrence per investigator's judgement, can be enrolled
* Had major surgery (example, major cardiopulmonary or abdominal operations) as per the investigator's judgment within 4 weeks before vaccination, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to participate in the study
* Has an acute illness (including acute respiratory illnesses) or body temperature of >=38.0 degree Celsius (ºC) (>=100.4 Fahrenheit [ºF ] within 24 hours prior to administration of study vaccine)
* Has had major psychiatric illness and/or drug or alcohol abuse which in the investigator's opinion would compromise the participant's safety and/or compliance with the study procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2192 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Cohort 2: Neutralizing Antibody Titers Against RSV A Strain as Measured by Virus Neutralizing Antibody (VNA) Assay | Day 15
  Neutralizing antibody titers against RSV A strain as measured by VNA Assay will be reported.
Cohort 1: Number of Participants with First Occurrence of Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) confirmed Respiratory Syncytial Virus (RSV) Mediated-lower Respiratory Tract Disease (LRTD) Over one RSV Season | Until end of RSV season (up to 11.5 months)
  Number of participants with first occurrence of RT-PCR confirmed RSV Mediated LRTD over one RSV season will be reported.

SECONDARY OUTCOMES:
Cohort 1 (Immuno Subset): Neutralizing Antibody Titers Against RSV A Strain | Day 1, 15, 85, and 169
  Neutralizing antibody titers against RSV A strain will be reported.
Cohort 1 (Immuno Subset) and 2: RSV A F protein in pre-fusion form Binding Antibodies as Assessed by Enzyme linked Immuno Sorbent Assay (ELISA) | Cohort 1: Day 1, 15, 85, and 169; Cohort 2: 14 days after vaccination (Day 15)
  Antibodies binding to RSV A F protein in pre-fusion form as assessed by ELISA will be reported
Cohorts 1 and 2: Number of Participants with Serious Adverse Events (SAEs) | Cohort 1: Up to 6 months after vaccination or end of RSV season, whichever comes later (up to 11.5 months); Cohort 2: Up to 6 months after vaccination
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Cohorts 1 and 2: Number of Participants with Adverse Events of Special Interest (AESIs) | Cohort 1: Up to 6 months after vaccination or end of RSV season, whichever comes later (up to 11.5 months); Cohort 2: Up to 6 months after vaccination
  Number of participants with AESIs will be reported. Thrombosis with thrombocytopenia syndrome is considered to be an AESI.
Cohort 1 (Safety Subset) and Cohort 2: Number of Participants with Solicited Systemic AEs After Vaccination | 7 Days after vaccination (Day 1 to Day 8)
  Solicited systemic AEs (fatigue, headache, myalgia, nausea and fever) will be noted in the participant diary for 7 days post-vaccination.
Cohort 1 (Safety Subset) and Cohort 2: Number of Participants with Solicited Local Adverse Events (AEs) After Vaccination | 7 Days after vaccination (Day 1 to Day 8)
  An AE is any untoward medical occurrence in a clinical study participant administered an investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. Solicited local AEs (including erythema, swelling, and pain/tenderness at the study vaccine injection site) will be noted in the participant diary for 7 days post-vaccination.
Cohort 1 (Safety Subset) and Cohort 2: Number of Participants with Unsolicited AEs After Vaccination | 28 days after vaccination (Day 1 to Day 29)
  Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Cohort 2: Neutralizing Antibody Titers Against RSV A Strain iso RSV A2 as Measured by VNA Assay in terms of Seroresponse rate | 14 days after vaccination (Day 15)
  Neutralizing antibody titers against RSV A strain as measured by VNA assay in terms of seroresponse rate will be reported. Seroresponse is defined as a 4-fold increase from baseline in Day 15 antibody titers.
Cohort 1: Number of Participants with First Occurrence of RT-PCR Confirmed RSV-mediated Acute Respiratory Infection (ARI) Over one RSV Season | Until end of RSV season (up to 11.5 months)
  Number of participants with first occurrence of any RT-PCR confirmed RSV-mediated ARI over one RSV season will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (30):
- Japan (30):
  - Shohokai Toda Internal Medicine and Neurology Clinic, Akashi-shi
  - Doujin Memorial Meiwa Hospital, Chiyoda-ku
  - Fukuwa Clinic, Chūō
  - Tokyo-Eki Center-Building Clinic, Chūōku
  - Tokyo Asbo Clinic, Chūōku
  - Tenjin Sogo Clinic, Fukuoka
  - Seikoukai New Medical Research System Clinic, Hachioji-shi
  - Hiroshima Station Clinic, Hiroshima
  - Medical Corporation JR Hiroshima Hospital, Hiroshima
  - Teine Keijinkai Hospital, Hokkaido
  - Aso Co.,Ltd Iizuka Hospital, Iizuka
  - Kishiwada Tokushukai Hospital, Kishiwada
  - Seikokai Omi Medical Center, Kusatsu-shi
  - Tohno Chuo Clinic, Mizunami-shi
  - Kojunkai Daido Hospital, Nagoya
  - Chubu Tokushukai Hospital, Nakagami-gun
  - Hanabusakai Shimamura Memorial Hospital, Nerima-ku
  - Yotsubashi Clinic, Osaka
  - Satou Hospital Miyagi, Osaki-shi
  - Jakushikai Banno Clinic, Ōta-ku
  - Keichikai Shimokitazawa Tomo Clinic, Setagaya-ku
  - Nanbu Tokushukai Hospital, Shimajiri-Gun
  - Clinical Research Hospital Tokyo, Shinjuku-ku
  - Ishinkai Oda Clinic, Shinjyuku-ku
  - Hanabusakai Shinei Clinic, Suginami-ku
  - Josuikai Olive Takamatsu Medical Clinic, Takamatsu
  - Ikebukuro Metropolitan Clinic, Tokyo-To
  - Kouwakai Kouwa Clinic, Toshima-ku
  - Senrichuo Ekimae Clinic, Toyonaka-shi
  - Tsuchiura Beryl Clinic, Tsuchiura-shi

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Tamura H, Momose A, Takato Y, Richuan Z, Bastian AR, Callendret B, Heijnen E. Phase 3 study of an Ad26.RSV.preF/RSV preF protein vaccine to evaluate the prevention efficacy of RSV-mediated lower tract disease, immunogenicity and safety in Japanese adults. Respir Investig. 2025 Jul;63(4):560-568. doi: 10.1016/j.resinv.2025.04.016. Epub 2025 May 3. PMID 40319702